CLINICAL TRIAL: NCT04362020
Title: Strategies to Maintain Radial Artery Patency Following Diagnostic Coronary Angiography - Subgroup of Patients on Oral Anticoagulants
Acronym: RAPID-2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Luebeck (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. Ingo Eitel, Director, University of Luebeck
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RAPID-2
Record Dates: First submitted 2020-04-22; First posted 2020-04-24 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Patient Undergoing Diagnostic Coronary Angiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group-1 (Experimental): No anticoagulation
  Interventions: Other: Distal radial access
- Group-2 (Active Comparator): ACT-guided anticoagulation
  Interventions: Other: Distal radial access

INTERVENTIONS:
Other: Distal radial access — Distal radial access and No anticoagulation
  Arms: Group-1
Other: Distal radial access — Distal radial access and ACT-guided anticoagulation
  Arms: Group-2

SUMMARY:
To investigate whether omitting systemic anticoagulation during transradial coronary angiography and/or a distal radial access reduce the risk of postprocedural radial artery occlusion

ELIGIBILITY:
Inclusion Criteria:

* Clinical indication to perform diagnostic coronary angiography
* Pretreatment with oral anticoagulants (phenprocoumon or direct oral anticoagulants [dabigatran, apixaban, rivaroxaban, or edoxaban])
* Age > 18 years
* Written informed consent

Exclusion Criteria:

* Already administered additional anticoagulation prior to coronary angiography
* Planned coronary intervention
* Preexisting radial artery occlusion or missing pulse at the potential puncture sites
* Allergy / intolerance to anticoagulants
* Active bleeding or comorbidity with elevated bleeding risk
* Pregnancy
* Inability to sign informed consent
* Participation in another trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2020-05-01 (Estimated); Primary Completion 2021-11-30 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Occurrence of postprocedural radial artery occlusion | Day 1
  Will be the occurrence of postprocedural radial artery occlusion assessed with high-resolution vascular ultrasound. Experienced sonographers will perform color Doppler ultrasound in all study patients after removal of the compression device to examine the radial, ulnar, and brachial arteries of the access forearm.

SECONDARY OUTCOMES:
Sonographic characteristics of radial artery occlusion | 3 Month
  Occlusion lengths or minimal residual perfusion

REFERENCES:
- [Derived] Stiermaier T, Grunewalder M, Patz T, Rawish E, Joost A, Meusel M, Marquetand C, Kurz T, Schmidt T, Frerker C, Fuernau G, Eitel I. Distal access and procedural anticoagulation to prevent radial artery occlusion after coronary angiography - the randomised RAPID trial. EuroIntervention. 2025 Apr 7;21(7):e366-e375. doi: 10.4244/EIJ-D-24-00846. PMID 40191883